CLINICAL TRIAL: NCT01478555
Title: A Dose-Finding Study To Compare The Safety, Tolerability, And Efficacy Of Differing Dosing Regimens Of ISV-101 (Bromfenac In DuraSite® Ophthalmic Solution) To Vehicle And DuraSite Alone In Dry Eye Disease Volunteers
Brief Title: A Dose-Finding Study Comparing InSite Vision, Inc. 101 to Vehicle and DuraSite Alone for Dry Eye Disease
Acronym: ISV-101
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Project postponed
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C-10-101-001
Record Dates: First submitted 2011-10-24; First posted 2011-11-23 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose 1 of Bromfenac in DuraSite (Experimental)
  Interventions: Drug: ISV 101
- Dose 2 of Bromfenac in DuraSite (Experimental)
  Interventions: Drug: ISV 101
- Dose 3 of Bromfenac in DuraSite (Experimental)
  Interventions: Drug: ISV 101
- DuraSite (Active Comparator)
  Interventions: Drug: ISV 101
- Vehicle (Active Comparator)
  Interventions: Drug: ISV 101

INTERVENTIONS:
Drug: ISV 101 — Bromfenac in DuraSite

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy in topical administration of differing dosing regimens of ISV-101 (Bromfenac in DuraSite® ophthalmic solution) compared to Vehicle and DuraSite alone.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers 18 years of age and older who have a diagnosis of moderate to severe dry eye disease.
2. Negative pregnancy test prior to the conduct of any protocol-specific procedure. The subject must use effective contraception for the duration of the study. Post menopausal is defined as having no menses for at least 12 consecutive months
3. Signature of the subject on the Informed Consent Form
4. Willing to avoid disallowed medication for the duration of the study.
5. Able to self-administer study drug (or have a caregiver available to instill all doses of study drug)
6. Able and willing to follow study instructions
7. Additional inclusion criteria also apply

Exclusion Criteria:

1. Females who are pregnant or nursing. Females of childbearing potential (not surgically sterilized or postmenopausal) may not participate in the study if they do not agree to use adequate birth control methods for the duration of the study).
2. Use of contact lenses during the study.
3. Use of any concomitant topical ocular medications except for artificial tears during the dosing period
4. Presence or history of treatment with systemic immunosuppressive or chemotherapeutic agents.
5. Prior or anticipated concurrent use of an investigational product or device that could confound the findings about Dry Eye in the study eye.
6. A condition or a situation, which in the investigator's opinion may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation
7. Known hypersensitivity to any component of the study drug or procedural medications
8. Participation in any other clinical trial within 30 days prior to screening
9. Known hypersensitivity to NSAIDS
10. Any active corneal epithelial/stromal pathology noted in the study eye at the screening visit
11. Any history of corneal surgery (including corneal crosslinking, radial keratotomy, corneal transplant, or LASIK)
12. Cataract surgery within the past year.
13. Known contraindication to the study drugs or any of their components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Corneal Fluorescein Staining | Week 8
Improvement in OSDI Scoring | Week 8